CLINICAL TRIAL: NCT05450731
Title: Effect of Cardiac Rehabilitation Exercise on the Recurrence of Atrial Fibrillation in Post-ablation Patients: a Randomized Controlled Pilot Study
Brief Title: Cardiac Rehab Post-atrial Fib Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/05/04
Record Dates: First submitted 2022-06-21; First posted 2022-07-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiac rehabilitation intervention group (Experimental): Participants assigned to the intervention group will participate in pre-post assessments and a 12-week supervised exercise based cardiac rehabilitation program at a designated local Pulse Heart Institute Cardiac Rehabilitation program.
  Interventions: Other: 12-week supervised exercise based cardiac rehabilitation program
- control group (No Intervention): Participants assigned to the control group will participate in pre-post assessments and will maintain usual care and current activity levels.

INTERVENTIONS:
Other: 12-week supervised exercise based cardiac rehabilitation program — 12-week exercise-based cardiac rehabilitation intervention on the recurrence of atrial fibrillation (AF) in patients at six- and twelve-months post-ablation procedure.
  Arms: cardiac rehabilitation intervention group

SUMMARY:
The aim of this study is to examine the effect of a 12-week exercise-based cardiac rehabilitation intervention on the recurrence of atrial fibrillation (AF) in patients at six- and twelve-months post-ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* ● Adult patients 18 years and older.

  * Willing to participate in the study after randomization to either an intervention group (cardiac rehabilitation exercise) or a control group (usual care).
  * Able to attend two pre and post study clinic visits at a local designated Pulse Heart Institute cardiac rehab program.
  * If randomized to the cardiac rehab intervention group can attend exercise rehab visits for 3 x per week for 12 weeks (36 visits) at a designated Pulse cardiac rehab program.
  * Has an active email address and phone number.
  * Documented diagnosis of Paroxysmal and persistent Atrial Fibrillation.
  * Undergone ablation treatment and is at a minimum of 2 weeks post ablation status.
  * Compliant with medication therapy including medications for heart rate control and anticoagulant(s).

Exclusion Criteria:

* ● Does not speak English.

  * Does not have clearance to participate in the study by their attending cardiologist.
  * Documented cardiovascular disease or pulmonary/respiratory disease that would qualify the patient for Cardiac, Pulmonary or Vascular Rehabilitation at a Pulse Heart Institute rehabilitation program.
  * Dementia or cognitive impairment.
  * Unable to participate in rehabilitation exercise due to physical limitations.
  * Greater than one prior ablation procedure
  * Long standing, chronic Atrial Fibrillation
  * Patients who have undergone posterior wall isolation ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to examine the effect of a 12-week exercise-based cardiac rehabilitation intervention on the recurrence of atrial fibrillation (AF) in 40 patients at six- and twelve-months post-ablation procedure. | 12 months after the first intake appointment
  Examine the effect of a 12-week exercise-based cardiac rehabilitation intervention on the recurrence of atrial fibrillation at 6- and 12-months post-ablation treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tacoma General Hospital, Tacoma, Washington, United States